CLINICAL TRIAL: NCT01247636
Title: Effect of Progressive Home-Exercise on Health-related Quality of Life, Balance and Mobility in Older People Discharge From an Outpatient Geriatric Clinic.
Brief Title: Home-Exercise vs General Physical Activity: Effect on Health-related Quality of Life
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Therese Brovold, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-03247
Record Dates: First submitted 2010-11-18; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2005-01

CONDITIONS: Health-Related Quality of Life
Keywords: HLRQ; Elderly; Balance; Mobility; Fear of falling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home-exercise (Experimental)
  Interventions: Other: Balance- training and home-exercise; Other: Balance-training and home-exercise

INTERVENTIONS:
Other: Balance- training and home-exercise — Balance-training admitted at the geriatric hospital Home-exercise or advice to be generally active
  Other Names: 1 intervention group; 1 control group
Other: Balance-training and home-exercise — The aim of the intervention was to enhance health-related quality of life, self-efficacy and physical function through education and exercise. The education program consisted of information given both oral and in writing regarding the benefits of physical activity. The aim was to increase the participants knowledge about the benefits of physical activity and to stimulate them to integrate physical activity into their immediate environment during daily routines. They were given an exercise-log and were advised to write down all their daily activities and exercise. The exercise program were conducted 2 times per week for 45 min per session. The content of these sessions were balance training with main focus on balance-exercises considered essential for daily living.
  Other Names: 1 home-exercise group; 1 activity group

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the effectiveness of an exercised-based programme developed for older people admitted at a geriatric outpatient clinic and to see if a home-exercise program enhances the effect. The outcomes considered is health-related quality of life, balance-self confidence, balance and mobility.

DETAILED DESCRIPTION:
Older people discharge from hospital often have decreased functional and physiological reserve that make them vulnerable of being dependent of others. Research have shown that older people discharge from hospital are vulnerable for functional decline during hospital stay and this decline can persist 6 to 18 months after discharge from hospital.Exercise interventions are proven to have effect on mobility, balance and falls among community-dwelling older people and several studies have shown that deconditioning as a consequence of disuse is reversible with training even in very old individuals. However, few studies have evaluated the effects of physical activity promotion and exercise intervention among elderly recently discharge from a geriatric outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* home-dwelling patients who were admitted at the geriatric clinic.
* Assessed by a doctor to tolerate training
* Able to walk in the corridor for 3 min with or without assistive device

Exclusion Criteria:

* Cognitive disorders mini mental status < 24

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | by the time of discharge mean 2 weeks after admission
Health-related quality of life | 3 months

SECONDARY OUTCOMES:
Functional balance (Berg Balance Scale) | by the time of discharge mean 2 weeks after admission and after 3 months
Functional mobility | by the time of discharge mean 2 weeks after admission, and after 3 months
  Timed up and go test and 6 min walk test
Functional strength | by the time of discharge mean 2 weeks after admission and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, Professor, Study Chair — No afflication
Locations (1):
- Ulleval University Hospital, Oslo, Oslo County, Norway